CLINICAL TRIAL: NCT01526304
Title: A Cross-Sectional Study To Investigate The Role Of FGF23, Klotho, And Sclerostin In Kidney Stone Formers
Brief Title: The Role Of FGF23, Klotho, And Sclerostin In Kidney Stone Formers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SFS
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — No intervention, only observational study

SUMMARY:
Kidney stones are very common in industrialized countries and the lifetime risk is about 10 to 15% in this population. Kidney stones are composed of inorganic and organic components. Calcium containing stones are the most common stone type accounting for more than 80% of kidney stones. Many factors predispose or contribute to the development of kidney stones, including genetic variants or mutations, diet, environmental factors, and behavior. To date, little is known on fibroblast growth factor (FGF23) levels in patients with calcium nephrolithiasis. FGF23 is crucial for phosphate homeostasis including physiological and pathophysiological conditions such as X-linked hypophosphatemic rickets and it seems that FGF23 is probably the most important regulator of serum phosphate and calcitriol (1,25(OH)2D3) levels in addition to parathyroid hormone (PTH) produced by the parathyroid gland. Novel factors such as Klotho and Sclerostin, which are involved in the bone-kidney-parathyroid endocrine axis, have been identified recently. Klotho is a putative aging suppressor gene and its deficiency results in osteopenia, hyperphosphaturia, and calcification. Klotho is mainly expressed in the kidney but also in the parathyroid gland and acts as a FGF23 specific co-receptor mediating FGF23 participation in the bone-kidney-parathyroid endocrine axis as described above. Sclerostin is a protein secreted by osteocytes that inhibits bone formation by osteoblasts. However, the potential role of FGF23, Klotho, and Sclerostin in nephrolithiasis is still poorly under-stood or even unexplored. The aim of this study is to test if levels of FGF23, Klotho, and Sclerostin are differentially regulated in kidney stone formers.

DETAILED DESCRIPTION:
Kidney stones are very common in industrialized countries and the lifetime risk is about 10 to 15% in this population. Men are more affected than women and the mean age of the patients is be-tween the fourth and sixth decade of life. Notably, a considerable percentage of patients experience recurrent kidney stones with a relapse rate of 50% in 5-10 years complicated by pain and urinary tract infections and potential loss of functional renal parenchyma with development of chronic renal failure in the long term. Kidney stones are composed of inorganic and organic components. Calcium containing stones are the most common stone type accounting for more than 80% of kidney stones. Many factors predispose or contribute to the development of kidney stones, including genetic variants or mutations, diet, environmental factors, and behavior. Among all factors, abnormal urinary pH and calcium excretion are predominant findings in stone formers and seem to play a major role in the pathogenesis of stone formation (1-5). Moreover, a significant percentage of patients with calcium nephrolithiasis and normal parathyroid function show hypophosphatemia and reduced renal phosphate reabsorption i.e. a renal phosphate leak (6-8) with resulting hyperphosphaturia. To date, little is known on fibroblast growth factor (FGF23) levels in patients with calcium nephrolithiasis (6). The authors demonstrated that FGF23 was increased in stone formers with renal phosphate leak when compared to controls. Also serum FGF23 concentration was strongly inversely associated with serum phosphate levels and rate of tubular phosphate re-absorption, respectively. This study suggests a role of FGF23 in the pathogenesis of calcium nephrolithiasis, however, more studies are necessary to confirm these findings. More, the influence of other novel factors involved in hyperphosphaturia has not been identified yet, such as Klotho.

FGF23 is crucial for phosphate homeostasis including physiological and pathophysiological conditions such as X-linked hypophosphatemic rickets and it seems that FGF23 is probably the most important regulator of serum phosphate and calcitriol (1,25(OH)2D3) levels in addition to parathyroid hormone (PTH) produced by the parathyroid gland (9-13). FGF23 is produced by osteocytes and osteoblasts, secreted in response to phosphate, and 1,25(OH)2D3, binds to the FGF receptor (FGFR)/Klotho complex, and acts as a phosphaturic hormone by reducing the expression of both sodium dependent phosphate cotransporters, namely NaPi2a and NaPi2c in renal proximal tubule cells (14). There is some evidence of PTH induced expression and secretion of FGF23 and on the other hand FGF23 decreases 1,25(OH)2D3 production and thus stimulates PTH production. In chronic kidney disease (CKD) patients, FGF23 is involved in CKD-related mineral and bone disorder (CKD-MBD) and has been shown to be an independent and probably more critical cardiovascular risk factor than phosphate (14).

Novel factors such as Klotho and Sclerostin, which are involved in the bone-kidney-parathyroid endocrine axis, have been identified recently. Klotho is a putative aging suppressor gene and its deficiency results in osteopenia, hyperphosphaturia, and calcification. Klotho is mainly expressed in the kidney but also in the parathyroid gland and acts as a FGF23 specific co-receptor mediating FGF23 participation in the bone-kidney-parathyroid endocrine axis as described above. Interestingly, secreted Klotho is also able to induce phosphaturia independently of FGF23 (15).

Sclerostin is a protein secreted by osteocytes that inhibits bone formation by osteoblasts. Deficiency of Sclerostin causes van Buchem disease and sclerosteosis, both rare sclerosing bone disorders, respectively. Interestingly, in humans, Sclerostin mRNA is expressed in several tissues, with high levels in the kidney whereas Sclerostin protein is only restricted to osteocytes. The exclusive effect of Sclerostin on bone formation and its deficiency causing bone disorders suggest a potential role of this molecule also in other diseases where bone homeostasis may be disarranged such as nephrolithiasis (16-18).

However, the potential role of FGF23, Klotho, and Sclerostin in nephrolithiasis is still poorly under-stood or even unexplored. The aim of this study is to test if levels of FGF23, Klotho, and Sclerostin are differentially regulated in kidney stone formers. Given the large number of kidney stone patients worldwide, the better understanding of the pathogenesis of kidney disease may provide the basis for the design of more individualized and specifically targeted therapeutics for this patient cohort.

ELIGIBILITY:
Inclusion criteria:

- stoneformer patients with signed informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stoneformer patients at the first outpatient stone clinic consultation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nilufar Mohebbi, MD, Principal Investigator — University Hospital Zurich, Division of Nephrology
Locations (1):
- University Hospital Zurich, Nephrology, Zurich, Canton of Zurich, Switzerland